CLINICAL TRIAL: NCT06884618
Title: A Phase I Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Clinical Activity of RO7673396 as a Single Agent and in Combination With Other Anticancer Therapies in Patients With Advanced Solid Tumors Harboring RAS Mutation(s)
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK) and Preliminary Clinical Activity of RO7673396 in Participants With Advanced Solid Tumors Harboring Rat Sarcoma Viral Oncogene Homolog (RAS) Mutation(s)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YO45758; 2024-519622-20-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-03-18; First posted 2025-03-19 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms
Keywords: RAS Mutated Solid Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stage I (Experimental): Participants with advanced solid tumors harboring RAS mutations will receive multiple ascending doses of RO7673396, as per a pre-defined dosing regimen until unacceptable toxicity or disease progression and/or loss of clinical benefit as determined by the investigator.
  Interventions: Drug: RO7673396
- Stage II (Experimental): Participants with advanced solid tumors harboring RAS mutations will receive RO7673396 at the dose determined in Stage 1, until unacceptable toxicity or disease progression and/or loss of clinical benefit as determined by the investigator.
  Interventions: Drug: RO7673396

INTERVENTIONS:
Drug: RO7673396 — RO7673396 will be administered as per the schedule specified in the protocol.

SUMMARY:
This study aims to evaluate the safety and tolerability of RO7673396 in participants with advanced solid tumors harboring RAS mutation(s). This study consists of two stages: Stage 1 (Dose Escalation) and Stage 2 (Dose Expansion). Stage 1 will define the recommended dose(s) for expansion (RDEs) of RO7673396. Stage 2 will evaluate preliminary anti-tumor activity of the RDE(s) defined in Stage 1 and of other doses of interest for future development in selected solid tumor indications.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented, locally advanced, recurrent, or metastatic incurable solid tumors
* Participants with measurable disease according to RECIST v1.1 assessed by the investigator
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy ≥12 weeks
* Adequate hematologic and end-organ function
* Confirmed presence of the RAS mutation(s)

Exclusion Criteria:

* Current participant or enrollment in another interventional clinical trial
* Known hypersensitivity or medical contraindication to any component of RO7673396 formulation
* Refractory nausea and vomiting, malabsorption, external biliary shunt, or significant small bowel resection that would preclude adequate study treatment absorption
* Known and untreated, or active central nervous system (CNS) metastases
* Participants with chronic diarrhea, short bowel syndrome or significant upper gastrointestinal (GI) surgery including gastric resection, a history of inflammatory bowel disease
* Treatment with chemotherapy, immunotherapy, biologic therapy, or an investigational agent as anti-cancer therapy within 4 weeks or five half-lives prior to initiation of study treatment
* Major surgical procedure within 28 days prior to initiation of study treatment, or incomplete recovery from surgery that would interfere with the determination of safety or efficacy of study treatment, or anticipation of need for a major surgical procedure during the study
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Known clinically significant liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-05-25 (Estimated)

PRIMARY OUTCOMES:
Stage I: Number of Participants With Adverse Events (AEs) | Up to approximately 40 months
Stage I: Number of Participants With Dose-limiting Toxicities (DLTs) | Up to Day 21
Stage II: Objective Response Rate (ORR) as Assessed by the Investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST V1.1) | Up to approximately 40 months

SECONDARY OUTCOMES:
Plasma Concentrations of RO7673396 and its Metabolite(s) | Up to approximately 49 months
Stage I: ORR as Assessed by the Investigator per RECIST V1.1 | Up to approximately 49 months
Stage I and II: Duration of Response (DOR) as Assessed by the Investigator per RECIST V1.1 | Up to approximately 49 months
Stage I and II: Progression-free Survival (PFS) as Assessed by the Investigator per RECIST V1.1 | Up to approximately 49 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- United States (6):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of Colorado - Anschutz Medical Campus - PPDS, Aurora, Colorado
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Florida Cancer Specialists - Sarasota (North Catttlemen Rd), Sarasota, Florida
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
- Australia (2):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Peter MacCallum Cancer Center, Parkville, Victoria
- Princess Margaret Hospital, Toronto, Ontario, Canada
- China (4):
  - Sun Yat-Sen University Cancer Center - Huangpu Campus, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center;Department of Thoracic Surgery, Guangzhou
  - Fudan University Shanghai Cancer Center, Shanghai
  - Hubei Cancer Hospital, Wuhan
- Prince of Wales Hospital, Hong Kong, Hong Kong
- New Zealand (2):
  - New Zealand Clinical Research - Auckland, Auckland
  - New Zealand Clinical Research - Christchurch, Christchurch
- National Cancer Centre - 30 Hospital Blvd, Singapore, Singapore
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing